CLINICAL TRIAL: NCT00690833
Title: Efficacy of Desonide (Desonatetm) Gel 0.05% in Younger and Older Subjects With Atopic Dermatitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wake Forest University (Other)
Responsible Party: Sponsor
Organization: Wake Forest University Health Sciences (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00002928; 32426
Record Dates: First submitted 2008-06-02; First posted 2008-06-05 (Estimated); Results first posted 2017-03-28 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- topical desonide hydrogel 0.05% (Experimental): Approximately 40 male and female subjects (about 20 age 3 months to <13 years and 20 age 13 and up) with mild to moderate atopic dermatitis will apply desonate gel twice daily to ATD
  Interventions: Drug: topical desonide hydrogel 0.05%

INTERVENTIONS:
Drug: topical desonide hydrogel 0.05% — apply the smallest amount of study medication possible that is just sufficient to cover all lesions of the standard cortisone-type medication twice daily (morning and evening) for up to 4 weeks to all of their AD lesions
  Other Names: Desonide gel

SUMMARY:
The purpose of this research study is to better understand how this study drug works when people use it to treat atopic dermatitis. Desonate has been approved by the US Food and Drug Administration (FDA) for atopic dermatitis.

DETAILED DESCRIPTION:
To assess the efficacy of a desonide hydrogel 0.05% in both young children (age <13) and older subjects (ages 13 and up) with mild to moderate atopic dermatitis

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 3 months or greater.
* Subjects must have diagnosis of mild to moderate atopic dermatitis by an investigator (a 2 or 3 on the IGA scale).
* Subjects must have >2% BSA involvement to be enrolled.
* Informed consent of participation must be given by parent or guardian if he or she is <7 years old. Children who are 7 to 18 years old will be given an assent form to sign.
* Moisturizers will be allowed during the study as long as the use remains stable from screening/baseline throughout the study.

Exclusion Criteria:

* Known allergy or sensitivity to topical desonide hydrogel in the subject.
* Inability to complete all study-related visits.
* Introduction of any other prescription medication, topical or systemic, for atopic dermatitis while participating in the study. Other than stable use of over the counter non-medicated moisturizers, all other topical treatments for AD must be stopped prior to study drug initiation. There will be no required washout for any topical therapies. Stable use of systemic therapies may be continued throughout the study.
* Requiring >130 gm of cream in a 4 week period.
* Pregnant women and women who are breastfeeding are to be excluded. Women of childbearing potential will be allowed to participate in the study, and these subjects will be required to use at least one form of birth control. Use of desonide in pregnant subjects is controversial and is only to be used when benefits outweigh the risks.

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2009-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Feldman, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences Dermatology, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Topical Desonide Hydrogel 0.05%
Started | 41
Completed | 39
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Topical Desonide Hydrogel 0.05%
Number analyzed (Participants) | 41
Age, Continuous [Median (Full Range); unit: years] | 13 [1 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 19
  White | 17
  More than one race | 2
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 41

OUTCOME MEASURES:

1. Primary Outcome: Investigator Global Assessment at Week 4
Description: The Investigator global assessment at Week 4 is based on an overall scale of 0-4 with 0 being clear and 4 being very severe
Time Frame: Week 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Topical Desonide Hydrogel 0.05%
Number analyzed (Participants) | 41
units on a scale | 2.3 (0.5)

ADVERSE EVENTS:
Arm/Group | Topical Desonide Hydrogel 0.05%
Serious Adverse Events (participants affected / at risk) | 0/41
Other Adverse Events (participants affected / at risk) | 0/41

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes